CLINICAL TRIAL: NCT01350206
Title: Hepatic Resection Versus Transcatheter Arterial Chemoembolization for Hepatocellular Carcinoma Complicated by Portal Vein Tumor Thrombosis.A Prospective and Randomized Clinical Trial
Brief Title: Hepatic Resection Versus Transcatheter Arterial Chemoembolization for Hepatocellular Carcinoma Complicated by Portal Vein Tumor Thrombosis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Cancer Center, Sun Yat-sen University, Cancer Center, Sun Yat-sen University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: HCC0011
Record Dates: First submitted 2011-05-06; First posted 2011-05-09 (Estimated); Last update posted 2011-05-09 (Estimated); Status verified 2010-04

CONDITIONS: Hepatocellular Carcinoma With PVTT
Keywords: Carcinoma,Hepatocellular; Liver Neoplasms; Therapeutic; Chemoembolization,; TACE; hepatic resection
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HR group (Experimental): HR was carried out under general anesthesia using a right subcostal incision with a midline extension. Intraoperative ultrasound was routinely performed. Pringle's maneuver was routinely used with a clamp/unclamp time of 10 minutes/5 minutes.Thrombectomy was performed according to the location and extent of PVTT. The en bloc technique was used for patients if the portal vein branch could be ligated with a sufficient safety margin between its root and the tip of the thrombus
  Interventions: Procedure: hepatic resection
- TACE group (Experimental): TACE with chemotherapy drugs (EADM 50mg, lobaplatin 50mg, and MMC 6mg )mixed with iodized oil lipidol
  Interventions: Procedure: TACE

INTERVENTIONS:
Procedure: hepatic resection — HR was carried out under general anesthesia using a right subcostal incision with a midline extension. Intraoperative ultrasound was routinely performed. Pringle's maneuver was routinely used with a clamp/unclamp time of 10 minutes/5 minutes.Thrombectomy was performed according to the location and extent of PVTT. The en bloc technique was used for patients if the portal vein branch could be ligated with a sufficient safety margin between its root and the tip of the thrombus
  Arms: HR group
Procedure: TACE — TACE with chemotherapy drugs (EADM 50mg, lobaplatin 50mg, and MMC 6mg )mixed with iodized oil lipidol
  Arms: TACE group

SUMMARY:
The treatment for Hepatocellular Carcinoma (HCC) with Portal Vein Tumor Thrombosis (PVTT) is still controversial, and there is no universally agreed protocol for its treatment. Transarterial chemoembolization (TACE) has become the most popular palliative treatment for patients with unresectable HCC, and it is no longer considered as a contraindication to HCC with PVTT. Unfortunately, the long term outcomes are generally poor for HCC treated with TACE, especially for HCC with PVTT. HR remains the only therapeutic option that may still offer a chance of cure. With advances in surgical techniques, it has become feasible to remove all gross tumors, including PVTT which has extended to the main portal vein, safely by surgery. This study aimed to evaluate the safety and efficacy of HR as compared with TACE to treat patients with HCC with PVTT. The investigators also aimed to identify patient groups that might benefit more from either treatment with HR or TACE.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is the sixth most common cancer and the third most frequent cause of cancer death worldwide. Hepatic resection (HR) is the conventional "curative" treatment for HCC. In both the European and the Unit States Proposed Guidelines for HCC, HR is recommended only for patients with preserved liver function and with a single HCC lesion. Unfortunately, because of tumor multifocality, portal vein invasion, and underlying advanced cirrhosis, only 10%-30% of HCCs are amenable to such a "curative" treatment at the time of diagnosis. Transarterial chemoembolization (TACE) has become the most popular palliative treatment for patients with unresectable HCC, and it is no longer considered as a contraindication to HCC with portal vein tumor thrombus (PVTT). Unfortunately, the long term outcomes are generally poor for HCC treated with TACE, especially for HCC with PVTT.

To improve on the results of treatment of HCC with PVTT, attempts have been made to perform HR for these patients . HCC with PVTT remains a contraindication to liver transplantation because of the high rate of tumor recurrence, and because of the severe shortage of donor organs. HR remains the only therapeutic option that may still offer a chance of cure. With advances in surgical techniques, it has become feasible to remove all gross tumors, including PVTT which has extended to the main portal vein, safely by surgery. More HCC with PVTT, which previously were considered as unresectable, have become resectable. Recent studies have even shown favorable long-term survival outcomes of HR in well-selected cases of HCC with PVTT. However, the survival outcomes of patients with HCC with PVTT treated with HR or with TACE have not been properly compared.

This study aimed to evaluate the safety and efficacy of HR as compared with TACE to treat patients with HCC with PVTT. The investigators also aimed to identify patient groups that might benefit more from either treatment with HR or TACE.

ELIGIBILITY:
Inclusion Criteria:

1. age between 18 and 75 years,
2. HCC with no previous treatment,
3. the presence of PVTT on imaging,
4. Eastern Co-operative Group performance status 0 ,
5. resectable disease, which is defined as the possibility of completely removing all gross tumors and retaining a sufficient liver remnant to sustain life, as assessed by our surgery team.

Exclusion Criteria:

1. the presence of extrahepatic spread on imaging,
2. a Child-Pugh class C liver cirrhosis, or ICG-R15 >30%, or evidence of hepatic decompensation including ascites, esophageal or gastric variceal bleeding or hepatic encephalopathy,
3. an American Society of Anesthesiologists (ASA) score ≥ 3

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2010-04; Primary Completion 2012-05 (Estimated); Study Completion 2013-05 (Estimated)

PRIMARY OUTCOMES:
overall survival | 1 year

SECONDARY OUTCOMES:
Time to progression | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: min-shan chen, Ph.D.,M.D., Principal Investigator — Cancer Center, Sun Yat-set University
Locations (1):
- Cancer Center Sun Yat-sen University, Guangzhou, Guangdong, China